CLINICAL TRIAL: NCT04309955
Title: Randomized Clinical Trial of Modified Versus Traditional Thoracic Drainage After Thoracoscopic Surgery for Lung Cancer
Brief Title: Modified Versus Traditional Thoracic Drainage After Thoracoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Kun Li, MD, Kun Li, MD, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kli3
Record Dates: First submitted 2020-03-08; First posted 2020-03-17 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Lung Neoplasms; Lung Cancer; Pulmonary Neoplasm; Postoperative Pain; Thoracoscopic Surgery
Keywords: chest tube; pigtail catheters; chest tube drainage; thoracic drainage; Lung Cancer; thoracoscopic surgery; Pulmonary Neoplasm
MeSH Terms: conditions — Lung Neoplasms; Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified thoracic drainage group (Experimental): After surgery, both a chest tube and a pigtail catheter are inserted into the middle and posterior axillary lines of the 7th intercostal space, respectively.
  Interventions: Procedure: pigtail catheter
- traditional thoracic drainage group (No Intervention): After surgery, only a chest tube is inserted into the midaxillary line of the 7th intercostal space, traditionally.

INTERVENTIONS:
Procedure: pigtail catheter — After inserting the chest tube, add a pigtail catheter into the posterior axillary lines of the 7th intercostal.
  Arms: modified thoracic drainage group

SUMMARY:
Lung cancer is the leading cause of cancer-related death worldwide. Thoracoscopic pulmonary resection is a prevalent management for early stage of lung cancer. Placement of traditional chest tube is the standard procedure after surgery, which causes pain that cannot be ignored. We aimed to determine whether a modified thoracic drainage strategy based on pigtail catheter associated with better clinical results compared with traditional methods after thoracoscopic surgery for lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18<age<80;
* Patients with lung cancer;
* Thoracoscopic lung resection;
* Single chest-tube insertion.

Exclusion Criteria:

* A history of preoperative chemotherapy or radiotherapy;
* Presence of distant tumor metastasis;
* Pneumonectomy;
* Dysfunction of cardiorespiratory system or other surgical contraindications.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Chest tube drainage duration | From date of operation until the date of chest tube removal, assessed up to 7 days
  The number of days from operation day to the day of chest tube removal
Volume of drainage | From date of operation until the date of removal of the chest tube and pigtail catheter, assessed up to 7 days.
  Total volume of thoracic drainage (ml)

SECONDARY OUTCOMES:
Postoperative hospital stay | From date of operation until the date of hospital discharge, assessed up to 30 days.
  The numbers of days of patients stay in the hospital after surgery

OTHER OUTCOMES:
Postoperative pain scores | Postoperative day 1, 2, 3, 4 and 5.
  Postoperative pain is evaluated by pain scores (0 [No pain] to 10 [Pain as bad as you can endure])

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Chongqing Municipality, China